CLINICAL TRIAL: NCT05603091
Title: Pressure Wave Guided Atrial Fibrillation Cryoablation: POLAR-WAVE Registry
Brief Title: Pressure Wave Guided Atrial Fibrillation Cryoablation
Acronym: POLAR-WAVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Adolfo Fontenla, Principal Investigator, Quirón Madrid University Hospital
Other Study IDs: POLAR-WAVE
Record Dates: First submitted 2022-10-20; First posted 2022-11-02 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Cryoablation; Pressure waveforms
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Pressure guided cryoablation: Patients undergoing cryoablation of atrial fibrillation with catheter-balloon, where the evaluation of the pulmonary veins occlusion will be assessed by the analysis of the pressure waveforms obtained from the tip of the catheter (without injecting contrast).
  Interventions: Procedure: cryoablation of pulmonary veins

INTERVENTIONS:
Procedure: cryoablation of pulmonary veins — Procedures are guided by pressure waveforms analysis, which are obtained by connecting the internal lumen of the catheter through the lateral port of the hemostatic valve attached to the catheter, to a pressure transducer connected in turn to a heparinized saline serum bag and to the cryoablation console.

SUMMARY:
Prospective multicenter observational study evaluating the performance of pressure wave-guided atrial fibrillation cryoablation used in accordance with clinical practice guidelines.

DETAILED DESCRIPTION:
The POLAR-WAVE registry is a prospective, multi-center, single-arm study evaluating the efficacy and safety of pressure-guided atrial fibrillation cryoablation, where the occlusion of pulmonary veins will be assessed by pressure waveforms (instead of contrast), over a follow-up period of 12 months.

This is a non-commercial, investigator-driven clinical study, coordinated by the main investigator from University Hospital "12th of October", Madrid, Spain. Several responsibilities are delegated to the Clinical Research Unit (University Hospital "12th of October", Madrid, Spain).

The study was planned according to the Good Clinical Practices. POLAR-WAVE Study has been approved by the Ethics Committee and Spanish Health Authorities. All participating patients must give written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Paroxysmal, persistent, or long-lasting persistent atrial fibrillation.
* Indication of pulmonary vein ablation according to clinical practice guidelines.

Exclusion Criteria:

* Previous ablation of atrial fibrillation.
* Thrombus in the left atrium.
* Rheumatic heart disease.
* Hypertrophic cardiomyopathy.
* Absolute contraindication to anticoagulation.
* Women in a state of pregnancy, lactation or childbearing age without contraception.
* Life expectancy < 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of patients who are candidates for paroxysmal or persistent AF ablation, in accordance with the conventional indications of the technique according to current European clinical practice guidelines
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Atrial tachycardia and/or atrial fibrillation (AT/AF) free survival | 12 months
  Proportion of patients without AT/AF episodes (excluding a window period of 3 months from ablation)

SECONDARY OUTCOMES:
Successfully completed ablation procedures | 12 months
  Proportion of pulmonary vein isolation (PVI) procedures exclusively guided by pressure
Symptoms associated with atrial fibrillation | 12 months
  European Heart Rhythm Association Symptom Scale (I-IV). Higher scores mean a worse outcome.
Safety events | 30 days
  Proportion of serious and non-serious procedure related events
Acute results of pressure guided cryoablation procedures (global and for each vein) | 1 day
  proportion of isolated veins, proportion of isolated veins with single application.
Performance of pressure guided cryoablation procedures | 1 day
  Total procedure time (min), dwell time in the left atrium (min), cryotherapy time (min), fluoroscopy time (min)
Temperature parameters obtained during pressure guided cryoablation procedures (global and for each vein) | 1 day
  * Minimum temperature (degrees Celsius)
  * Temperature at 30 seconds (degrees Celsius)
  * Temperature at 60 seconds (degrees Celsius)
Time parameters obtained during pressure guided cryoablation | 1 day
  * Time up to -40 degrees Celsius (sec)
  * Time up to -50 degrees Celsius (sec)
  * Defrosting time up to 0 degrees Celsius (sec)
  * Defrosting time up to +15 degrees Celsius (sec)
Radiation dose | 1 day
  Mean radiation required for pulmonary vein isolation (Gycm2)

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Fontenla, MD, PhD, Study Chair — Hospital Universitario 12 de Octubre, Madrid. Spain
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Background] Siklody CH, Minners J, Allgeier M, Allgeier HJ, Jander N, Keyl C, Weber R, Schiebeling-Romer J, Kalusche D, Arentz T. Pressure-guided cryoballoon isolation of the pulmonary veins for the treatment of paroxysmal atrial fibrillation. J Cardiovasc Electrophysiol. 2010 Feb;21(2):120-5. doi: 10.1111/j.1540-8167.2009.01600.x. Epub 2009 Sep 28. PMID 19793145
- [Background] Raizada A, Gedela M, Shaikh KA, Apte N, DeHaan M, Stanton C. Pressure-Guided cryoablation of pulmonary veins in atrial fibrillation: A fast and effective strategy. Indian Heart J. 2017 Mar-Apr;69(2):223-225. doi: 10.1016/j.ihj.2016.11.330. Epub 2016 Dec 5. PMID 28460771
- [Background] Hasegawa K, Miyazaki S, Kaseno K, Hisazaki K, Amaya N, Miyahara K, Aiki T, Ishikawa E, Mukai M, Matsui A, Aoyama D, Shiomi Y, Tama N, Ikeda H, Fukuoka Y, Morishita T, Ishida K, Uzui H, Tada H. Pressure-guided second-generation cryoballoon pulmonary vein isolation: Prospective comparison of the procedural and clinical outcomes with the conventional strategy. J Cardiovasc Electrophysiol. 2019 Oct;30(10):1841-1847. doi: 10.1111/jce.14080. Epub 2019 Aug 4. PMID 31328311
- [Background] Heeger CH, Pott A, Sohns C, Riesinger L, Sommer P, Gasperetti A, Tondo C, Fassini G, Moser F, Lucas P, Weinmann K, Bohnen JE, Dahme T, Rillig A, Kuck KH, Wakili R, Metzner A, Tilz RR. Novel cryoballoon ablation system for pulmonary vein isolation: multicenter assessment of efficacy and safety-ANTARCTICA study. Europace. 2022 Dec 9;24(12):1917-1925. doi: 10.1093/europace/euac148. PMID 36026521
- [Background] Martin A, Fowler M, Breskovic T, Ouss A, Dekker L, Yap SC, Bhagwandien R, Albrecht EM, Cielen N, Richards E, Tran BC, Lever N, Anic A. Novel cryoballoon to isolate pulmonary veins in patients with paroxysmal atrial fibrillation: long-term outcomes in a multicentre clinical study. J Interv Card Electrophysiol. 2022 Dec;65(3):609-616. doi: 10.1007/s10840-022-01200-5. Epub 2022 Apr 12. PMID 35412168
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916